CLINICAL TRIAL: NCT03734107
Title: Improving Health Communication During the Transition From Pediatric to Adult Diabetes Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Randi Streisand, Principal Investigator, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30004426
Record Dates: First submitted 2018-11-01; First posted 2018-11-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: transition to adult medical care; adolescents and young adults; health communication; adherence; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to the intervention group or standard care comparison group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREP-DC Intervention (Experimental): 50 participants will be randomized to the Plan, Reflect, and Engage with Providers for Diabetes Care (PREP-DC) intervention. Participants will complete 3 intervention sessions with study interventionists and will receive text messages and other study resources during the active intervention period (3 months).
  Interventions: Behavioral: Plan, Reflect, and Engage with Providers for Diabetes Care
- Standard Care Comparison (No Intervention): 50 participants will be randomized to standard care and will participate in regular diabetes clinic visits and receive standard materials on the transition to adult diabetes care, as they would have done without participation in this study.

INTERVENTIONS:
Behavioral: Plan, Reflect, and Engage with Providers for Diabetes Care — Behavioral intervention designed to improve health communication skills and readiness for adult diabetes care
  Other Names: PREP-DC
  Arms: PREP-DC Intervention

SUMMARY:
Adolescents and young adults (AYAs; ages 17-23) with type 1 diabetes are at high risk for negative health outcomes, including poor glycemic control and disengagement from the health care system. The deterioration of glycemic control occurs in parallel with the assumption of independent self-care skills and preparation for adult diabetes care. Effective communication between AYAs and health care providers may be a critical contributor to diabetes self-care skills during the transition to adult diabetes care and related glycemic control. This research will attempt to better prepare adolescents and young adults for adult diabetes care by delivering innovative intervention content focused on both health communication skills and transition readiness skills. The investigators aim to leverage innovative technologies to improve developmentally-appropriate communication skills related to planning for clinic visits, disclosing and discussing diabetes-related concerns, and optimizing glucose data review in preparation for adult diabetes care. Adolescents and young adults with type 1 diabetes (ages 17-23) who are planning to transition to adult diabetes care within the next 6-8 months will be enrolled in the study and randomized to either the intervention group or a standard care control group. Medical, communication and psychosocial data (including A1c, glucose monitoring frequency, communication quality, health care engagement, depressive symptoms) will be collected from adolescent and young adult participants and health care providers at baseline and two follow-up time points, approximately 4 months post-baseline and approximately 8-12 months post-baseline after the transfer to adult diabetes care. This intervention has the potential to improve diabetes self-care skills, including engagement with health care providers, and glycemic control in AYAs with type 1 diabetes during the vulnerable period of transfer to adult diabetes care. The results of this work will inform best practices for the transition to adult diabetes care and can be translated into clinical care.

DETAILED DESCRIPTION:
Research Design and Methods Overview of Study Design & Procedure. The aim of this randomized controlled trial (RCT) is to determine the efficacy of a behavioral intervention targeting health communication skills and diabetes self-management skills in preparation for the transfer to adult diabetes care, compared to usual care. The intervention, Plan, Reflect, and Engage with Providers for Diabetes Care (PREP-DC), consists of three intervention sessions with a study interventionist, paired text messages, and access to glucose management software. It is expected that adolescents and young adults allocated to the intervention condition (PREP-DC) will evidence: 1) better glycemic control (lower A1c); 2) shorter gap in time between the last visit in pediatric diabetes care and the first visit in adult diabetes care; 3) better diabetes management (better adherence to the diabetes regimen); 4) fewer reported complications (e.g. hospitalizations and emergency department visits). A total of 100 adolescent and young adult participants (ages 17-23) will be randomly allocated in a 1:1 ratio to either the PREP-DC intervention condition (n=50) or usual care (n=50; standard care comparison condition): all participants receive standard resources for transition to adult diabetes care as part of usual care in both conditions.

Participants include 100 adolescents and young adults (ages 17-23) diagnosed with T1D for at least one year (anticipated 50% female) seen for diabetes care at Children's National Medical Center (CNMC) in Washington, DC. Eligible participants will self-identify as planning to transfer to adult diabetes care within the upcoming 6-8 months. Participants in the PREP-DC intervention will complete three intervention sessions with study team members over a 3 month period (approximately 1 intervention session per month). Two sessions will be with a trained study interventionist focusing on communication with health care providers and preparation for medical visits and adult diabetes care. One session will be with a certified diabetes education focusing on problem-solving using glucose data and glucose data review. PREP-DC intervention participants will also receive text messages (3-4 messages/week) for the 3 month intervention period supporting intervention content. Participants also will be given information about accessing glucose management software specific to their diabetes devices and related study resources (e.g. study website). Participants are evaluated at baseline (pre-randomization to intervention or standard care comparison group) and follow-up (approximately 4 months post-baseline and approximately 8-12 months post-baseline after the transition to adult diabetes care).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type1 diabetes for ≥ 1 year
* Able to adequately understand, speak, and read English to benefit from participation
* Ready and consistent text messaging access to participate
* Within 6-8 months of planned transfer to adult diabetes care

Exclusion Criteria:

* Other life-threatening disease (e.g. cancer) or major psychiatric disorder (e.g. schizophrenia) that significantly limits participation
* Pervasive developmental disorder that significantly limits participation

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 8 months post-baseline
  measurement of hemoglobin A1c (A1c; reported as a percentage)
Number of days to first adult diabetes care visit | 8 months post-baseline
  Number of days between the last visit in pediatric diabetes care and the first visit in adult diabetes care (reported as number of days)
Adherence to the diabetes care regimen | 8 months post-baseline
  Participant report on the Diabetes Management Questionnaire (DMQ), a self-report measure of adherence to the diabetes care regimen. The DMQ consists of 20 items scored on a 0-4 Likert Scale. The measure has a total score; the mean score on all items is calculated and multiplied by 25 to arrive at the total score (possible range 0-100). A higher score indicates greater adherence to diabetes management.
Diabetes-related hospitalizations | 8 months post-baseline
  Participant report and medical record review of reported diabetes-related hospitalizations for the duration of the study period. The total number of hospitalizations is summed.

CONTACTS AND LOCATIONS:
Overall Officials: Randi Streisand, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States